CLINICAL TRIAL: NCT00675090
Title: A Single Blind, Placebo-controlled, Randomised Study in Mild to Moderate Alzheimer's Disease Patients to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK239512, a Selective Histamine H3 Receptor Antagonist
Brief Title: Bridging Study With GSK239512 In Patients With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H3B109689
Record Dates: First submitted 2008-04-24; First posted 2008-05-08 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — GSK239512

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK239512 (Experimental): GSK239512 oral tablets
  Interventions: Drug: GSK239512
- Placebo (Placebo Comparator): Placebo to match tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK239512 — GSK239512 oral tablets once a day
  Arms: GSK239512
Drug: Placebo — Placebo tablets to match once a day
  Arms: Placebo

SUMMARY:
This is a safety and tolerability study to investigate the effect of GSK239512 on mild to moderate Alzheimers disease patients. The dose of GSK239512 will be titrated to reach the most well tolerated dose in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a clinical diagnosis of probable Alzheimer's disease
* The subject has an MMSE score at screening of 12 to 26 for Part A and 16-26 for Part B.
* Age ≥ 50 and above.
* If female, the subject must be post-menopausal (i.e. 12 months without menstrual period) or surgically sterile.
* Male subjects must be willing to abstain from sexual intercourse with pregnant or lactating women; or be willing to use a condom/spermicide in addition to having their female partner use another form of contraception if the woman could become pregnant, from the time of the first dose of GSK239512 until 84 days following completion of the study.
* The subject has the ability to comply with the study procedures.
* The subject has a permanent caregiver and is willing to attend all study visits for Parts A and B.
* The subject has provided full written informed consent prior to the performance of any protocol specific procedure, or if unable to provide informed consent due to cognitive status, full written informed consent on behalf of the subject has been provided by a legally acceptable representative.
* The caregiver has provided his / her written consent prior to the performance of any protocol specific procedure.

Exclusion Criteria:

* In the opinion of the investigator, following review of CT/MRI scans in the past 12 months and completion of neurological review there could be other probable causes of dementia
* History of significant psychiatric illness such as schizophrenia or bipolar affective disorder that in the opinion of the Investigator would interfere with participation in the study, or current depression (a score of ≥8 on the Cornell Scale for Depression in Dementia), or subjects with other psychiatric features in their AD which would in the opinion of the investigator, would increase risk to safety.
* History of significant sleep disturbance, for example, when it is associated with nocturnal wandering, nocturnal confusion / disorientation / agitation, which in the opinion of the investigator, may increase safety risk.
* History or presence of known or suspected seizures, unexplained significant loss of consciousness within last 6 months. Subjects who had febrile seizures in childhood may be included if these ceased by age 10 and they have had no other type of seizure in their medical history and have not been on anti-epileptic medications.
* History or presence of significant cardiovascular, gastro-intestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, or any other clinically relevant abnormality, medical or psychiatric condition, which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* History of alcohol or other substance abuse, according to the Diagnostic and Statistical Manual of Mental Disorders - Substance related disorders (DSM-IV) criteria.
* Clinically significant abnormalities in laboratory tests, including subjects with active liver disease or uncontrolled thyroid disease.
* Uncontrolled hypertension with systolic BP ≥160 and/or diastolic ≥95 mmHg. Subjects with controlled hypertension with systolic BP < 160 mmHg and diastolic <95 mmHg for at least 4 weeks are acceptable.
* Systolic BP <100 mmHg and/or diastolic <60 mmHg.
* Subjects with ECG criteria outside ranges specified in the protocol
* History of hypersensitivity to GSK239512 or its excipients.
* Treatment with cholinesterase inhibitors, (including Tacrine), memantine or selegiline within the previous month. No patients with AD who are already on these medications at the time of screening will be recruited, as it would be unethical to withdraw these medications for study participation. Only AD subjects who are not yet on these medications, or who have withdrawn from these medications for other reasons previously, may be enrolled into this study.
* Subjects who are currently taking or who have taken in the last month anti-psychotic drugs (typical or atypical dopaminergic antagonists or modulators) or mood stabilization drugs (including SSRI, DNRI, SNRI, MAO inhibitors, tricyclic antidepressants, lithium, valproate, carbamazepine).
* Subjects who are currently taking Pgp inhibitors or any CYP3A4 inhibitors.
* Subjects on chronic sedative medications (≥ 4 days per week for the past 4 weeks).
* Subject or caregiver is an immediate family member or employee of the participating Investigator, any of the participating site staff or GSK staff.
* Has received any other investigational treatment in the previous 3 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-02-21 (Actual); Primary Completion 2009-06-16 (Actual); Study Completion 2009-06-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by adverse events, vital signs clinical laboratory measurements and validated clinical assessment scales. | Days 8, 15, 22 and 29

SECONDARY OUTCOMES:
Pharmacodynamics measured by computerized cognitive tests and validated clinical rating scales. Also investigating the Pharmacokineticsat trough concentrations (Cmin) after GSK239512 repeat dosing on days 8, 15, 22 and 29 and 15. | days 8, 15, 22 and 29

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Australia (2):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Heidelberg Heights, Victoria
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, Seoul, South Korea
- United Kingdom (3):
  - GSK Investigational Site, Cambridgeshire, Cambridgeshire
  - GSK Investigational Site, London
  - GSK Investigational Site, Southall

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nathan PJ, Boardley R, Scott N, Berges A, Maruff P, Sivananthan T, Upton N, Lowy MT, Nestor PJ, Lai R. The safety, tolerability, pharmacokinetics and cognitive effects of GSK239512, a selective histamine H(3) receptor antagonist in patients with mild to moderate Alzheimer's disease: a preliminary investigation. Curr Alzheimer Res. 2013 Mar;10(3):240-51. doi: 10.2174/1567205011310030003. PMID 23521503
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study H3B109689 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/H3B109689?search=study&study_ids=H3B109689#rs
- Available data/document: Dataset Specification: H3B109689 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: H3B109689 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: H3B109689 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: H3B109689 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: H3B109689 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: H3B109689 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: H3B109689 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register